CLINICAL TRIAL: NCT00005003
Title: Mapping the Genetic Component of Hand-Use Preference
Brief Title: Genetic Component of Handedness
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000094; 00-C-0094
Record Dates: First submitted 2000-03-23; First posted 2000-03-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-04

CONDITIONS: Healthy
Keywords: Handedness; Laterality; Linkage; VNTR/Dinucleotide; Dinucleotide; High-Frequency-Trait Analysis

SUMMARY:
Some functions are generally controlled by the right side of the brain and others by the left. One of the most easily observed examples of this "lateral specialization" of the brain is handedness-that is, a person's preference for using either the right or the left hand. This study will try to determine how the genetic component of handedness is inherited. It will test the theory that a single gene is involved in determining handedness and will try to locate the gene.

Families with at least two left-handed siblings aged eight years or older and at least one right-handed parent are eligible to participate in this study.

The left-handed siblings and both parents will fill out a brief questionnaire on hand usage, obtain a tissue sample taken from inside the cheek, and return the questionnaire and the sample by mail to the study researchers. The tissue sample will be used for DNA gene mapping.

Participants will be given a kit and instructions for obtaining the sample, along with mailing envelopes. Cheek swab sampling basically involves using a small brush to gently brush a layer of cells off of the inner wall of the cheek and then dropping the brush tip into a preservative.

The information gained from this study may provide insight into aspects of brain development that can be of medical benefit in the future.

DETAILED DESCRIPTION:
The purpose of this protocol, based on the hypothesis that human hand-use preference (handedness) is largely dependent on the action of a single locus, is to collect samples allowing us to map a "handedness gene" via detection of linkage to any of eight potential candidate genes/regions or via a whole or partial genome scan. We calculate that a full 300 marker genome scan of 100 parents and sibling pairs (allowing linkage analysis at 10 cM resolution), or the equivalent amount of data from partial scans of 300 families, has a high likelihood of allowing us to map the proposed gene. Eligible families, consisting of pairs of left-handed siblings plus at least one right-handed parent, were identified during Phase I of this study in 1996-1998, with approval from the now-lapsed FCRDC IRB. In Phase II of this study, we have collected cheek swab samples for DNA isolation from members of 100 eligible families for use in the mapping studies. DNA samples will not be linked back to individuals but grouped under a random family code that links to a database with limited information, including hand use preference and family structure. In the next phase, we wish to map the locus from cheek swab samples we have on hand.

ELIGIBILITY:
INCLUSION CRITERIA:

Members of families meeting the following criteria are eligible to participate:

Have two left-handed siblings.

Have at least one right-handed parent with no other known left-handed first degree relatives.

EXCLUSION CRITERIA:

All members of a family may be excluded if the right-handed parents or the left-handed siblings will not participate.

Individuals in families whose left-handed siblings are under the age of eight are not eligible to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400
Dates: Start 2000-03; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Corballis MC. The genetics and evolution of handedness. Psychol Rev. 1997 Oct;104(4):714-27. doi: 10.1037/0033-295x.104.4.714. PMID 9337630
- [Background] Dellatolas G, Luciani S, Castresana A, Remy C, Jallon P, Laplane D, Bancaud J. Pathological left-handedness. Left-handedness correlatives in adult epileptics. Brain. 1993 Dec;116 ( Pt 6):1565-74. doi: 10.1093/brain/116.6.1565. PMID 8293288
- [Background] Levin M, Nascone N. Two molecular models of initial left-right asymmetry generation. Med Hypotheses. 1997 Nov;49(5):429-35. doi: 10.1016/s0306-9877(97)90092-x. PMID 9421811